CLINICAL TRIAL: NCT05560022
Title: Study of the Total Hip Prosthesis With a HYPE Stem in Hip Arthroplasty
Brief Title: Prospective and Obsevational Study of Total Hip Prothesis: HYPE Stem
Status: Active, not recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-01-NH-HYPE-Novae
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Hip Arthropathy
Keywords: Total Hip Prothesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to validate the performance and the safety of the HYPE (SERF) prothesis in compliance with the 93/42/EEC directive and in relation to the recommendations of the MEDDEV 2.7.1 guide ( guideline for post-market follow-up), which provides for the implementation of a systematic procedure for the follow-up of clinical data in order to verify the performance claimed for medical devices .

ELIGIBILITY:
Inclusion Criteria:

* Man or women
* Degenerative or inflammatory hip pathology requiring a total hip replacement
* Primary or secondary osteoarthritis
* Advanced joint destruction resulting from rhumatoid arthritis or traumatic arthritis
* Fracture or avascular necrosis
* Sub-capital fracture and displaced transcervical as well as for bone defects stages I to IIb of PAPROSKY
* Traumatic joint destruction
* Following previous intervention, provided that the new device does not interfere with the material in place (osteosynthesis, joint reconstruction, arthrodesis, hemi-arthroplasty, total arthroplasty

Exclusion Criteria:

* People with diminished mental faculties
* Known current pregnancy
* Breast-feeding
* Neurological disorders or other pathologies that may influence locomotion
* Septic antecedent on hip to operate
* Patient requiring a bone graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The implantation of the total hip prothesis will be performed in patients with a hip pathology in the first intention or during total prothesis revision
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2031-01-20 (Estimated); Study Completion 2031-01-20 (Estimated)

PRIMARY OUTCOMES:
Assess the Survival rate to Total Hip Prothesis combining a HYPE stem and a SERF cup in hip replacements | per operative period to 10 years
  Survival according to Kaplan Meier

SECONDARY OUTCOMES:
Assess the improvement in PMA scores and HHS score as well as patient satisfaction | per operative period to 10 years
Adverse events | per operative period to 10 years
  Type and occurrence of adverse events
Patient satisfaction | per operative period to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de ROUEN, Rouen, France